CLINICAL TRIAL: NCT02095808
Title: Metabolic Biomarkers in Thoracic Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kemp Kernstine, PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU 052012-065
Record Dates: First submitted 2013-04-17; First posted 2014-03-26 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Surgery (Experimental): The 13C-glucose solution will be given intravenously. It will be started at about the same time as the start of surgery, according to the study guidelines.
  The 13C-glucose IV solution will be stopped once the surgeon has removed the tumor tissue.
  Interventions: Procedure: Imaging Biomarkers

INTERVENTIONS:
Procedure: Imaging Biomarkers — Want to see if using 13C-glucose helps in detecting cancer and deciding on a treatment plan.

SUMMARY:
The purpose of this research study is to develop a method of using magnetic resonance imaging (MRI) to evaluate lung tumors and other thoracic malignancies. An MRI is a scanning device that uses magnets to make images (pictures) of the body. This study is being done to determine what series of reactions (metabolic pathways) pulmonary nodules use as they burn sugar as fuel for growth. The manner in which the tumor burns (metabolizes) sugar for fuel is being investigated by using a natural, slightly modified, sugar solution (13C-glucose) and studying a small sample of the tumor once it is removed at the time of surgery.

DETAILED DESCRIPTION:
The recent report of the findings of the National Lung Screening Trial indicates that screening a high-risk population using low dose CT results in a 20% reduction in lung cancer mortality. At our institution, some of positive nodules that are 1 cm or larger would be imaged using combined fluoro-deoxyglucose positron emission tomography (FDG PET)/CT. Highly suspicious nodules would be biopsied if the risks were manageable. Otherwise, the suspicious nodules not eligible for biopsy and so-called "indeterminate" nodules are followed using CT to be evaluated for interval growth.

The overall goal of this project is to assess several very promising imaging biomarkers that can reflect either the physiological or metabolic status of these nodules in order to develop more accurate imaging algorithms for follow-up that are either less invasive or do not use ionizing radiation or both. Based on our experience with other cancers and our preliminary results in lung cancer, we have identified four potential imaging studies that we believe have the potential to result in validated "imaging biomarkers" that can either individually, or in combination, characterize malignancies. Since tumors tend to exhibit angiogenesis and altered vascular permeability, we and others, have found that analyses of dynamic contrast enhanced MRI (DCEMRI) can be employed as "imaging biomarkers" for malignancy. Tumors often exhibit higher cellularity than benign or normal tissue suggesting that pixel-by-pixel ADC values derived from diffusion weighted MRI could be useful imaging biomarkers. Finally, measuring alterations in metabolic fluxes through the use of pathway specific C-13 labeled compounds, a technique pioneered here at the Advanced Imaging Research Center (AIRC) at UT Southwestern, has shown the capability of providing metabolic fingerprints for malignant and benign tissue. This approach, while invasive, could identify and validate markers that can be detected non-invasively in future studies. We will also employ advanced metabolomics methods to identify potential signature "onco-metabolites" in these lung cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have known or probable malignant lesions requiring surgical biopsy or excision.
2. Subjects of all races and ethnic origins over 18 years of age.

Exclusion Criteria:

1. Not a surgical candidate.
2. Poorly controlled diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-03-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
DCE-MRI | One time - within 5 days of the scheduled surgery
  Physicians and researchers will review the results of the imaging to determine if the patient will receive the [U-13C] glucose infusion.

SECONDARY OUTCOMES:
C-13 isotopomer | During the infusion period blood samples will be collected every 30 minutes (for 2-3 hours) until the end of tumor sampling for mass spec and NMR analyisis of C-glucose in the blood.
  Employ C-13 isotopomer analysis and metabolomics on specimens obtained from resected tissue of suitable patients in this cohort to determine the metabolic alterations present in lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Kemp H Kernstine, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States